CLINICAL TRIAL: NCT02100865
Title: Solar Powered Oxygen Delivery: An Open-label Non-inferiority Comparison to Standard Oxygen Delivery Using Oxygen Cylinders
Brief Title: Solar Powered Oxygen Delivery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0206-01
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Pneumonia; Hypoxemia
MeSH Terms: conditions — Pneumonia; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solar powered oxygen (Experimental): Solar panels used to drive an oxygen concentrator to deliver at stream of oxygen at approximately 90% FiO2 and a rate of 1-5L/min.
  Interventions: Device: Solar powered oxygen
- Oxygen from cylinders (Active Comparator): Conventional oxygen delivery from compressed gas cylinders
  Interventions: Device: Oxygen from cylinders

INTERVENTIONS:
Device: Solar powered oxygen
  Arms: Solar powered oxygen
Device: Oxygen from cylinders
  Arms: Oxygen from cylinders

SUMMARY:
Globally, approximately 2.1 million children die of pneumonia each year. Most deaths occur in resource-poor settings in Africa and Asia. Oxygen (O2) therapy is essential to support life in these patients. Large gaps remain in the case management of children presenting to African hospitals with respiratory distress, including essential supportive therapies such as supplemental oxygen. We hypothesize that a novel strategy for oxygen delivery, solar-powered oxygen, can be implemented in remote locations and will be non-inferior to standard oxygen delivery by compressed gas cylinders.

DETAILED DESCRIPTION:
Arterial hypoxemia in pneumonia results from several mechanisms: pulmonary arterial blood flow to consolidated lung resulting in an intrapulmonary shunt, intrapulmonary oxygen consumption, and ventilation-perfusion mismatch. Hypoxemia is a risk factor for mortality in pediatric pneumonia, and was associated with a 5-fold increased risk of death in studies from Kenya and Gambia.

In one report from Nepal, the prevalence of hypoxemia (SpO2 < 90%) in 150 children with pneumonia was 39% overall, with increasing rates of hypoxemia across strata of pneumonia severity (100% of very severe, 80% of severe and 17% of pneumonia patients). General features of respiratory distress were associated with hypoxemia in this study, including chest indrawing, lethargy, grunting, nasal flaring, cyanosis, inability to breastfeed or drink.

Few studies have reported on the use of solar powered oxygen (SPO2) delivery. One online report describes the use of a battery-powered oxygenator in the Gambia that could be adapted to use solar power (http://www.dulas.org.uk). Otherwise, our intervention is to our knowledge the first example of SPO2 delivery.

New ways to deliver oxygen for children with pneumonia in Africa could improve outcomes and save numerous lives. If this study documents the non-inferiority of SPO2 relative to standard oxygen delivery, this novel method of providing life-saving oxygen could be rolled out across centres in sub-Saharan Africa where oxygen cylinders are not widely available and electrical power is not reliable. The potential energy efficiency, low cost and ease of use make solar power an attractive avenue of investigation for use in resource-constrained settings. Proof-of-concept that the sun can be used to drive oxygen delivery could stimulate commercial interest in this technology. The SPO2 system could thus achieve rapid penetration into the most remote or rural settings in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Age <13 years
* IMCI defined pneumonia, severe pneumonia or very severe disease
* Hypoxemia (SpO2<90%) based on non-invasive pulse oximetry
* Hospital admission warranted based on clinician judgment
* Consent to blood sampling and data collection

Exclusion Criteria:

* SpO2 ≥90%
* Suspected pulmonary tuberculosis
* Outpatient management
* Denial of consent to participate in study

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Until end of hospitalization (usually 3 to 7 days)
  The number of days from admission to discharge. Criteria for discharge are standardized and are assessed daily.

SECONDARY OUTCOMES:
Mortality | At hospital discharge (usually 3 to 7 days)
  In-hospital mortality will be quantified.
Duration of supplemental oxygen therapy | Until hospital discharge (usually 3 to 7 days)
  Time to wean patient off oxygen. This is assessed daily using standard procedures.
Proportion of patients successfully oxygenated | 6 hours
  Success defined as achieving a post-oxygen saturation above 90% within 6 hours.
Oxygen delivery system failure | During hospitalization (usually 3 to 7 days)
  Failure defined as need for backup oxygen to maintain SpO2>90%.
Cost | Until hospital discharge (usually 3 to 7 days)
  Cost of oxygen cylinders (control arm) and cost of equipment (capital investment - solar oxygen intervention arm).
Lambaréné Organ Dysfunction Score (LODS) | Until hospital discharge (usually 3 to 7 days)
  This simple published clinical score predicts mortality in children with malaria, but may also have prognostic value in pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Hawkes, MD, PhD, Principal Investigator — University of Alberta; Robert O Opoka, MBChB, MPH, Principal Investigator — Makerere University
Locations (1):
- Jinja Regional Referral Hospital, Jinja, Uganda

REFERENCES:
- [Result] Duke T, Wandi F, Jonathan M, Matai S, Kaupa M, Saavu M, Subhi R, Peel D. Improved oxygen systems for childhood pneumonia: a multihospital effectiveness study in Papua New Guinea. Lancet. 2008 Oct 11;372(9646):1328-33. doi: 10.1016/S0140-6736(08)61164-2. Epub 2008 Aug 15. PMID 18708248
- [Derived] Hawkes MT, Conroy AL, Namasopo S, Bhargava R, Kain KC, Mian Q, Opoka RO. Solar-Powered Oxygen Delivery in Low-Resource Settings: A Randomized Clinical Noninferiority Trial. JAMA Pediatr. 2018 Jul 1;172(7):694-696. doi: 10.1001/jamapediatrics.2018.0228. PMID 29800014
- [Derived] Nyende S, Conroy A, Opoka RO, Namasopo S, Kain KC, Mpimbaza A, Bhargava R, Hawkes M. Solar-powered oxygen delivery: study protocol for a randomized controlled trial. Trials. 2015 Jul 9;16:297. doi: 10.1186/s13063-015-0814-y. PMID 26156116
- See also: Global Health Uganda is the non-governmental organization (NGO) partner in Uganda — http://globalhealthuganda.org/